CLINICAL TRIAL: NCT05449444
Title: A 24-week, Multicenter, Randomized, Double Blind, Placebo-controlled, Dose-range Finding Phase II Study to Compare Efficacy and Safety of Oral Masitinib to Placebo in Treatment of Patients With Severe Mast Cell Activation Syndrome (MCAS) With Handicap Unresponsive to Optimal Symptomatic Treatment
Brief Title: Masitinib for the Treatment of Severe Mast Cell Activation Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AB20006; 2021-005406-96 (EudraCT Number)
Record Dates: First submitted 2022-07-02; First posted 2022-07-08 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Mast Cell Activation Syndrome
MeSH Terms: conditions — Mast Cell Activation Syndrome | interventions — masitinib

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel-group, multicenter comparative study with ascending dose titrations of masitinib and matching placebo
Who Masked: Participant, Investigator
Masking Description: Eligible patients will be randomized by means of a computerized central randomization system called IWRS (interactive web response system).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Masitinib (4.5) & BSC (Experimental): Masitinib 4.5 mg/kg/day administered as an add-on to optimal concomitant symptomatic treatment (i.e. best supportive care, BSC). Participants receive masitinib (3.0 mg/kg/day) for 4 weeks, given orally twice daily, with a dose escalation to 4.5 mg/kg/day for the remainder of the treatment period. Each ascending dose titration is subjected to a safety control.
  Interventions: Drug: Masitinib 4.5 mg/kg/day; Other: Best supportive care
- Masitinib (6.0) & BSC (Experimental): Masitinib 6.0 mg/kg/day administered as an add-on to optimal concomitant symptomatic treatment (i.e. best supportive care, BSC). Participants receive masitinib (3.0 mg/kg/day) for 4 weeks, given orally twice daily, with a dose escalation to 4.5 mg/kg/day for4 weeks of treatment, then a second dose escalation to 6 mg/kg/day for the remainder of the treatment period. Each ascending dose titration is subjected to a safety control.
  Interventions: Other: Best supportive care; Drug: Masitinib 6.0 mg/kg/day
- Placebo & BSC (Placebo Comparator): Placebo administered as an add-on to optimal concomitant symptomatic treatment (i.e. best supportive care, BSC). Participants receive a matched dose placebo, given orally twice daily.
  Interventions: Drug: Placebo; Other: Best supportive care

INTERVENTIONS:
Drug: Masitinib 4.5 mg/kg/day — Masitinib 4.5 mg/kg/day
  Other Names: AB1010
  Arms: Masitinib (4.5) & BSC
Drug: Placebo — Matching placebo
  Other Names: Placebo Oral Tablet
  Arms: Placebo & BSC
Other: Best supportive care — Optimal concomitant symptomatic treatments. Includes: H1- and H2-antihistamines, sodium cromoglicate, antidepressants, antileukotrienes, proton pump inhibitors, and corticosteroids.
  Other Names: BSC
Drug: Masitinib 6.0 mg/kg/day — Masitinib 6.0 mg/kg/day
  Other Names: AB1010
  Arms: Masitinib (6.0) & BSC

SUMMARY:
To evaluate the efficacy and safety of two dosing schemes of oral masitinib versus matching placebo in the treatment of patients suffering from severe MCAS with handicap unresponsive to optimal symptomatic treatment.

DETAILED DESCRIPTION:
Multicenter, double-blind, placebo-controlled trial comparing two different dosing schemes over a 24-week treatment period.

Dosing scheme #1: Oral masitinib treatment at 3 mg/kg/day for 4 weeks, then a switch to 4.5 mg/kg/day for the remainder of the treatment period, versus placebo with a matching titration scheme. Randomization 2: 1 (Masitinib MCAS: Placebo MCAS).

Dosing scheme #2: Oral masitinib treatment at 3 mg/kg/day for 4 weeks, then a switch to 4.5 mg/kg/day for 4 weeks, then a second switch to 6 mg/kg/day for the remainder of the treatment period versus placebo treatment with a matching titration scheme. Randomization 2: 1 (Masitinib MCAS: Placebo MCAS)

ELIGIBILITY:
Inclusion Criteria include:

* Patient with mast cell activation syndrome (MCAS).
* Patient with severe symptoms over the 14-day run-in period defined as at least one of the following: Pruritus score ≥ 9; Number of flushes per week ≥ 8; Hamilton rating scale for depression (HAMD-17) score ≥ 19
* Patient with documented treatment failures of his/her handicap(s) (within last two years) with at least two of the symptomatic treatments used at optimized dose.
* Patients must be on a stable dose of Anti-H1 for a minimum of 4 weeks before screening and should remain at a stable dose throughout the study period.

Exclusion Criteria include:

* Previous treatment with any Tyrosine Kinase Inhibitor.
* Any change in the symptomatic treatment of MCAS, including systemic corticosteroids, or administration of any new treatment for MCAS within 4 weeks prior to screening.
* Patient with systemic indolent mastocytosis.
* Female patients who are pregnant or are breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Confirmed response at 50% | 24 weeks
  Confirmed response at 50%, defined as an improvement with respect to the baseline values of 50% for Pruritus, Flushes and Depression (HAMD-17 score) which should be confirmed from the previous visit.
  Handicaps at baseline defined as: pruritus score ≥ 9; number of flushes per week ≥ 8; HAMD-17 score ≥ 19.

SECONDARY OUTCOMES:
Cumulative response | week 8 to week 24
  Cumulative (every patient visit) response at 75% on 3 handicaps (pruritus, flush, depression) from week 8 to week 24. Analysis will be performed using Generalized Estimating Equations (GEE) model with stratification.
Confirmed response (75%) | 24 weeks
  Confirmed response at 75%, defined as an an improvement with respect to the baseline values of 75% for Pruritus, Flushes and Depression (Hamilton Depression Rating Scale) which should be confirmed from the previous visit. The Hamilton Depression Rating Scale (HAMD-17) has 17 items and is scored between 0 and 4 points. Scores of 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression; the maximum score being 52.
Patient-Reported Outcome for Symptom Severity (PROSS) | 24 weeks
  Changes in MCAS symptom severity will also be assessed using the Patient-Reported Outcome for Symptom Severity (PROSS) questionnaire. Total and individual symptom scores will be determined at baseline and at every visit until Week 24.The PROSS questionnaire has 11 items and is scored between 0 and 10 points. A score of 0 is an absence of the symptom and a score of 10 is very severe; the maximum score being 110.

CONTACTS AND LOCATIONS:
Overall Officials: Julien Rossignol, MD, Principal Investigator — Reference Centre for Mastocytosis (CEREMAST), Necker Hospital, Paris, France
Locations (4):
- St Charles Clinical Research, Weldon Spring, Missouri, United States
- France (3):
  - Centre Hospitalier Universitaire Amiens-Picardie, Amiens
  - Necker-Enfants Malades Hospital, Centre de référence des Mastocytoses (CEREMAST), Paris
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No
No Masitinib is under clinical investigation and has not yet been approved in any sought-after indication by any health authority worldwide. As such, there is no plan for data-sharing at this point in time.

REFERENCES:
- [Background] Lortholary O, Chandesris MO, Bulai Livideanu C, Paul C, Guillet G, Jassem E, Niedoszytko M, Barete S, Verstovsek S, Grattan C, Damaj G, Canioni D, Fraitag S, Lhermitte L, Georgin Lavialle S, Frenzel L, Afrin LB, Hanssens K, Agopian J, Gaillard R, Kinet JP, Auclair C, Mansfield C, Moussy A, Dubreuil P, Hermine O. Masitinib for treatment of severely symptomatic indolent systemic mastocytosis: a randomised, placebo-controlled, phase 3 study. Lancet. 2017 Feb 11;389(10069):612-620. doi: 10.1016/S0140-6736(16)31403-9. Epub 2017 Jan 7. PMID 28069279
- [Derived] Latham BD, Oskin DS, Crouch RD, Vergne MJ, Jackson KD. Cytochromes P450 2C8 and 3A Catalyze the Metabolic Activation of the Tyrosine Kinase Inhibitor Masitinib. Chem Res Toxicol. 2022 Sep 19;35(9):1467-1481. doi: 10.1021/acs.chemrestox.2c00057. Epub 2022 Sep 1. PMID 36048877